CLINICAL TRIAL: NCT03687307
Title: What Are the Three Dimensional Soft Tissue Changes That Occur After Orthognathic Surgery for Skeletal Class II Patients? Pre-test Post-test Quasi Experimental Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Moussa, Assistant lecturer, Cairo University
Other Study IDs: cebd-cu-2017-04-05
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Orthognathic Surgery
Keywords: class II,; soft tissue changes; CBCT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of the study is to establish reference data that could be used for the creation of more accurate three dimensional prediction of soft tissue outcome.

DETAILED DESCRIPTION:
in this study, 15 skeletal class 2 orthognathic patients will be selected. CBCT and proface will be done preoperatively. after the surgery and 6 months later the imaging investigations will be repeated to investigate the soft tissue changes that have resulted due to the bone movement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class II skeletal deformity
* Patients must be over 18 years of age to allow for growth cessation
* Patients must not have any systemic condition which contraindicates general anaesthesia

Exclusion Criteria:

* o patients with cleft palate

  * patients with syndromes affecting their craniofacial structure
  * patients with facial scars
  * patients with severe facial asymmetry

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with class 2 skeletal deformity, over 18 years and younger than 40
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
3D soft-tissue changes (linear) | 6 months
  the changes that have occurred in the soft tissue of the face after undergoing orthognathic surgery

SECONDARY OUTCOMES:
Proportion of soft tissue change to hard tissue change | 6 months
  the distance that the soft tissue has moved compared to the underlying bone, as a percentage.
Is the esthetic outcome as expected/imagined? | 6 months
  using a 100mm visual analogue scale the patient will be asked to score how the aesthetic outcome measured against his expectations. 0mm is the worst score where the changes havent met the expectations at all and 100mm is where the outcome has perfectly met the expectation.
3D soft-tissue changes (angular) | 6 months
  the changes that have occurred in the soft tissue of the face after undergoing orthognathic surgery
3D soft-tissue changes (volumetric) | 6 months
  the changes that have occurred in the soft tissue of the face after undergoing orthognathic surgery

IPD SHARING:
Plan to Share IPD: Yes